CLINICAL TRIAL: NCT01173627
Title: An Open-Label, Randomized, Two-Period, Crossover Study to Evaluate the Bioequivalence of an Oral Transmucosal Test Troche Formulation of Fentanyl Citrate (400 mcg) Compared to an Equivalent Dose of a Commercially Available Reference Drug Product (Actiq 400 mcg, Cephalon, Inc.) in Normal Human Subjects Under Fasting Conditions
Brief Title: Bioequivalence of a Test Troche Formulation of Fentanyl Citrate (400 mcg) Compared to Actiq® 400 mcg, Cephalon, Inc.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Herbert Neuman, MD/Chief Medical Officer, Mallinckrodt
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 9204-06-840
Record Dates: First submitted 2010-07-29; First posted 2010-08-02 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Pain
Keywords: Bioequivalence; Fentanyl
MeSH Terms: conditions — Pain | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A - Test fentanyl citrate 400 mcg troche (Experimental): Test fentanyl citrate 400 mcg troche
  Interventions: Drug: Test fentanyl citrate 400 mcg troche
- B - Actiq 400 mcg (Active Comparator): Actiq 400 mcg
  Interventions: Drug: Actiq 400 mcg

INTERVENTIONS:
Drug: Test fentanyl citrate 400 mcg troche — Test fentanyl citrate 400 mcg troche administered as a single dose under fasted conditions
  Arms: A - Test fentanyl citrate 400 mcg troche
Drug: Actiq 400 mcg — Actiq 400 mcg administered as a single dose under fasted conditions
  Arms: B - Actiq 400 mcg

SUMMARY:
The purpose of this study was to evaluate the oral bioequivalence of the Mallinckrodt test fentanyl citrate oral transmucosal 400 mcg troche compared to Actiq 400 mcg (Cephalon, Inc.) under fasting conditions.

DETAILED DESCRIPTION:
Fentanyl is an opioid analgesic with pharmacological effects similar to morphine. Fentanyl interacts predominately with the opioid µ-receptor. In clinical settings, fentanyl exerts its principal pharmacologic effects on the central nervous system. The fentanyl citrate oral transmucosal troche, Actiq (Cephalon, Inc.), is indicated only for the management of breakthrough cancer pain in patients with malignancies who are already receiving and who are tolerant to prior therapy for their underlying persistent cancer pain.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant, non-lactating females, 18 years of age or older with a minimum body weight of 120 pounds and a body mass index (BMI) between 19 and 29 inclusive.
* Female subjects must be postmenopausal for at least one year, surgically sterile, or using a reliable method of contraception (oral, transdermal, or injectable hormonal contraceptive; condom with spermicide; IUD; abstinence, etc.) for at least 30 days prior to and for the duration of study participation.
* Normal, healthy status confirmed by required screening assessments.
* Subjects must be able to provide written consent and agree to abide by the study requirements.
* Subjects must be able to demonstrate they understand and can perform the dosing procedure correctly using a placebo troche at check-in to Period 1.

Exclusion Criteria:

* If female, a positive pregnancy test at any time during the study, pregnant, lactating, or likely to become pregnant during the study.
* Female subjects of childbearing potential who have not used adequate forms of birth control within 30 days of dosing.
* History of conditions that might contraindicate or require caution be used in the administration of fentanyl or naltrexone, including: renal impairment, hepatobiliary or pancreatic disease, gastrointestinal obstruction, cardiac disease, obstructive pulmonary disease, acute or severe bronchial asthma, hypercarbia, elevated intracranial pressure, depleted blood volume, paralytic ileus, or hypersensitivity or idiosyncratic reaction to fentanyl, naltrexone, or any opioids.
* History of any drug allergy, hypersensitivity, or intolerance which would compromise the safety of the subject or the study.
* History of chronic alcohol, drug, or narcotic abuse, chronic use of tranquilizers, sedatives, aspirin, antibiotics, or other medications.
* History of malignancy, stroke, or diabetes; cardiac, renal, liver, and pulmonary disease.
* History of anxiety, tension, severe agitation, psychiatric disorders, psychosis, or mental depression requiring hospitalization, psychotherapy, and/or medication.
* History or diagnosis of epilepsy or other seizure disorder.
* History of abdominal and/or pelvic surgery within the last 5 years, except elective surgical sterilization.
* History of acute abdominal conditions or gastrointestinal disease including, but not limited to, peptic ulcer, diverticulitis, bowel obstructions, adhesions, ileus, gastritis, and chronic diarrhea.
* Subjects presenting with acute illness.
* Administration of any other investigational drug during the 30 days prior to study entry.
* Subjects who have smoked or used nicotine-containing products within 6 months prior to study entry.
* Donation or significant loss of whole blood (480 mL or more) within 30 days or plasma within 14 days prior to study entry, including that withdrawn during the conduct of any other clinical study.
* Positive test results for HIV, hepatitis B, or hepatitis C.
* Positive test results for drugs of abuse or alcohol.
* Subjects who have taken prescription drugs, except hormonal contraception, within 14 days or over-the-counter medications (including herbal preparations) within 7 days prior to study drug administration except for standard daily dose multivitamins, which are excluded after check-in to Period 2.
* Any subject experiencing adverse events to the -13 and/or -1 hour doses of naltrexone, that in the investigator's opinion, are indicative of possible previous opioid use/abuse, or that would prevent tolerance of additional doses of naltrexone, will be withdrawn from the study prior to dosing with fentanyl.
* Subjects with dental braces or partial dentures.
* Subjects presenting with a history of gum disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-08; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Average bioequivalence is established if the 90% confidence interval on the ratio of formulation averages for AUCt, AUCinf, and Cmax are contained in the interval [80%, 125%]. | 30 hours

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Neuman, MD, Study Director — Mallinckrodt
Locations (1):
- PRACS Institute, Ltd, Fargo, North Dakota, United States